CLINICAL TRIAL: NCT00675480
Title: Aspiration Thrombectomy as an Adjunctive Therapy to Primary Angioplasty in Patients With ST Segment Elevation Myocardial Infarction
Brief Title: Thrombectomy in Acute Myocardial Infarction
Acronym: TAMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Michał Ciszewski, MD, PhD, Institute of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2PO5C00527
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Acute Myocardial Infarction
Keywords: myocardial infarction, thrombectomy, salvage index
MeSH Terms: conditions — Myocardial Infarction | interventions — Thrombectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- T (Experimental): Patients treated with thrombectomy: T
  Interventions: Procedure: Thrombectomy
- P (Active Comparator): Patients treated with standard PCI with stent implantation
  Interventions: Procedure: Primary angioplasty

INTERVENTIONS:
Procedure: Thrombectomy — Aspiration Thrombectomy prior to stent implantation in patients with ST segment elevation myocardial infarction
  Other Names: Rescue (Boston Scientific); Diver (Invatec)
  Arms: T
Procedure: Primary angioplasty — Standard primary angioplasty with stent implantation
  Other Names: Bare metal stent implanted during primary angioplasty
  Arms: P

SUMMARY:
The purpose of the study is to determine whether thrombus removal with aspiration thrombectomy for acute myocardial infarction reduces the infarct size.

DETAILED DESCRIPTION:
Acute myocardial infarction is caused by an abrupt occlusion of coronary vessel or severe reduction of coronary flow. It has been shown that the reperfusion therapy significantly improves the clinical outcome. Currently the optimal strategy is the primary angioplasty with stent implantation. The treatment is recommended by AHA/ACC and ESC if can be performed within 90 minutes from the first medical contact. However there is still a certain percentage of procedure failure. To further improve the outcome new techniques and devices are tested . Aspiration thrombectomy may facilitate the reperfusion by reducing thrombus burden. The aim of the study is to assess if adjunctive thrombectomy may improve clinical outcome in patients with an acute ST segment elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

1. First acute myocardial infarction with ST segment elevation within 12 hours from pain onset
2. Culprit lesion in left anterior descending or right coronary artery.
3. Coronary flow assessed in TIMI scale ≤ 2
4. Presence of total coronary occlusion or angiographically visible thrombus in the culprit vessel
5. Patient signed informed consent

Exclusion Criteria:

1. Cardiogenic shock.
2. Culprit lesion in left circumflex coronary artery.
3. Status post coronary artery by-pass grafting
4. Previous myocardial infarction
5. Status post percutaneous coronary intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2004-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Myocardial salvage index assessed with SPECT MIBI. | 5-8 days

SECONDARY OUTCOMES:
In hospital mortality | in hospital, before discharge
ST segment resolution after PCI; | 90 minutes
CK-MB AUC | 72 hours
Corrected TIMI frame count | immediately post PCI

CONTACTS AND LOCATIONS:
Overall Officials: Michal Ciszewski, MD, PhD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, Warsaw, Poland

REFERENCES:
- [Derived] Ciszewski M, Pregowski J, Teresinska A, Karcz M, Kalinczuk L, Pracon R, Witkowski A, Ruzyllo W. Aspiration coronary thrombectomy for acute myocardial infarction increases myocardial salvage: single center randomized study. Catheter Cardiovasc Interv. 2011 Oct 1;78(4):523-31. doi: 10.1002/ccd.22933. Epub 2011 Jun 6. PMID 21234920